CLINICAL TRIAL: NCT06004583
Title: Relationships Between Disease Severity and The C-Reactive Protein/Albumin Ratio and Various Hematological Parameters in Patients With Acne Vulgaris
Brief Title: C-Reactive Protein/Albumin Ratio and Acne Vulgaris
Status: Completed | Type: Observational
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Erdal Pala, Ass.Prof, Ataturk University
Other Study IDs: 30.12.2021/567
Record Dates: First submitted 2023-08-16; First posted 2023-08-22 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Acne Vulgaris
Keywords: acne vulgaris; CRP albumin ratio
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Acne group: Acne Vulgaris Diagnosed Patients
  Interventions: Diagnostic Test: Biochemical blood analysis
- Control group: Healthy participants
  Interventions: Diagnostic Test: Biochemical blood analysis

INTERVENTIONS:
Diagnostic Test: Biochemical blood analysis — Serum CRP and albumin levels

SUMMARY:
Objective: Acne vulgaris, an inflammatory disease, was investigated in this study with the claim that C-reactive protein (CRP) / albumin ratio and some hematological parameter ratios have the potential to be used as inflammatory markers to monitor disease severity and prognosis.

Methods: A descriptive cross-sectional study was conducted with two groups of patients aged 18-65 years, 61 patients diagnosed with acne vulgaris and 35 healthy control patients, and routine hemogram and biochemical parameters were compared. The Global Acne Severity Index was used to determine the severity of acne vulgaris.

ELIGIBILITY:
Inclusion Criteria:

* Acne vulgaris patients diagnosed by a dermatologist
* Healthy participants without acne
* 18-40 years of age
* Voluntary participation

Exclusion Criteria:

* Aged below18 or above 40 years
* Not voluntarily participated patents
* Pregnants, breast milked mothers, emergency situations

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Acne vulgaris patients and control healthy individuals
Sampling Method: Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2022-01-05 (Actual); Primary Completion 2023-02-02 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
CRP/albumin ratio | 3 months
  Statistical difference between groups

SECONDARY OUTCOMES:
Usage of CRP/albumin ratio as a Biomarker | 3 months
  New detection of CRP/albumin ratio as a new biomarker in the Acne patients

CONTACTS AND LOCATIONS:
Locations (1):
- AtaturkU, Erzurum, Turkey (Türkiye)